CLINICAL TRIAL: NCT00781287
Title: Impact of Raltegravir (Isentress/MK-0518) - Containing Regimens on HIV-1 Infected CD4+ T-Cells During Acute and Early HIV-1 Infection: A Randomized, Controlled Study Comparing Standard Antiretroviral Therapy to Standard Therapy Plus Raltegravir
Brief Title: Raltegravir (Isentress/MK-0518) and HIV-1 Infected CD4 Cells During Acute/Early HIV-1
Acronym: UW PIC 330
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment too slow.
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ann Collier, Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34908-D
Record Dates: First submitted 2008-10-24; First posted 2008-10-28 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: human immunodeficiency virus; raltegravir; primary HIV infection; HIV-1
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltegravir + 3-drug anti-HIV therapy (Experimental)
  Interventions: Drug: 3-drug anti-HIV therapy; Drug: Raltegravir
- 3-drug anti-HIV therapy (Active Comparator)
  Interventions: Drug: 3-drug anti-HIV therapy

INTERVENTIONS:
Drug: 3-drug anti-HIV therapy — 3 FDA-approved drugs, including two nucleos(t)ide reverse transcriptase inhibitors and either a non-nucleoside reverse transcriptase inhibitor or a protease inhibitor (Low dose ritonavir can be used to enhance the protease inhibitor and is not considered one of the 3 anti-HIV drugs)
Drug: Raltegravir — 400 mg BID PO
  Other Names: Isentress
  Arms: Raltegravir + 3-drug anti-HIV therapy

SUMMARY:
This is an investigator-initiated, two-year, randomized, controlled, single-center, open-label, pilot study comparing 3-drug highly active antiretroviral therapy (HAART) to 3-drug HAART plus raltegravir for persons with acute and early HIV-1 infection. The study will test the hypothesis that use of the integrase inhibitor raltegravir (400 mg BID orally) to inhibit the integration step of the HIV-1 life cycle in conjunction with HAART in subjects with recently acquired HIV-1 infection will decrease the number of HIV-1 infected CD4+ T-cells to a greater extent than a 3-drug HAART regimen.

DETAILED DESCRIPTION:
The study will be conducted at the UW Primary Infection Clinic and the UW AIDS Clinical Trials Unit. Secondary objectives will characterize safety, tolerability, plasma HIV-1 RNA and CD4+ T-cell values. The 3-drug HAART will be chosen and provided by the subject.

ELIGIBILITY:
Inclusion Criteria:

* Acute or Early HIV-1 infection
* HIV-1 RNA > or equal to 500 copies/mL
* Acceptable safety lab results (specified in protocol)
* Negative pregnancy test for females
* Willingness to use contraception (for females of reproductive potential

Exclusion Criteria:

* Prior receipt of investigational HIV-1 vaccine
* Use of immunomodulators other than systemic steroids within 30 days before entry
* Serious medical or psychiatric illness that would interfere with study participation
* Active drug or alcohol use that would interfere with study participation
* Allergy/hypersensitivity to raltegravir
* Pre- or Post-exposure prophylaxis for the exposure that led to HIV-1 acquisition
* Pregnancy or breastfeeding
* History of malignancy (other than localized squamous cell or basal cell cancer of the skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2012-02 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Number of HIV-1 infected CD4+ T-cells measured by a quantitative HIV-1 DNA PCR assay | 96 weeks

SECONDARY OUTCOMES:
CD4+ T-cells | 96 weeks
Plasma HIV-1 RNA | 96 weeks
Grade 3 and 4 signs and symptoms or laboratory toxicities at least one grade higher than baseline | From study drug start to 8 weeks after drug discontinuation
Plasma HIV-1 RNA | Baseline to Week 8
Tolerability (Discontinuation of raltegravir) | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ann C. Collier, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Primary Infection Clinic, Seattle, Washington, United States